CLINICAL TRIAL: NCT03266263
Title: Improving Education of Community Chain of Survival Through Innovative Teaching, Implementing Teamwork Skills, and Survey on Attitude and Willingness: A Pilot Study
Brief Title: A Study of Improving Education of Community Chain of Survival
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201606085RIND
Record Dates: First submitted 2017-08-17; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2016-08

CONDITIONS: Cardiac Arrest Circulatory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- automatic computer-led feedback (Experimental): automated feedback for CPR quality provided by computers
  Interventions: Device: automatic computer-led feedback
- instructor-led feedback (Active Comparator): feedback for CPR quality provided by instructors
  Interventions: Other: instructor-led feedback

INTERVENTIONS:
Device: automatic computer-led feedback — automated feedback software for CPR quality, including compression depth, rate, recoil, hands-off time, and ventilation volume
  Arms: automatic computer-led feedback
Other: instructor-led feedback — feedback for CPR quality by instructors
  Arms: instructor-led feedback

SUMMARY:
"High-quality cardiopulmonary resuscitation (CPR)" and "early defibrillation" are the most important parts of "the chain of survival", and they are highly associated with the survival rate and life quality of patients with cardiac arrest. It needs the witness to perform bystander CPR and use the automated external defibrillator (AED) if CPR and defibrillation are expected to be performed earlier. Nevertheless, few patients with cardiac arrest received bystander CPR in Taiwan. It might be caused by some reasons. First, traditional training programs were inefficient and ineffective in the retention of skills and thus students were not confident in their CPR skills after receiving training programs. Second, the current training module focused on personal skill training only and lacked teamwork skills training. It led to poor performance of the students in actual resuscitation scene, where on-scene resuscitators were usually more than one. Third, the current training contents did not improve the attitudes and willingness of performing bystander CPR and it caused people who had received training program did not resuscitate the patients finally. To improve the above-mentioned problem, a three-year research project will be implemented. The aims of the project are the following:

1. to explore the effect of different teaching contents and hand-on practice feedback methods on the students' performance of chest compressing, ventilating and using AED in the CPR and AED training courses.
2. to analyze the current situation of teamwork when CPR and AED were performed, to build up the collaborating module accordingly and evaluate the effect of the new module on the students' performance of chest compressing, ventilating and using AED after the module is introduced into the training course.
3. to understand the factors affecting the motivations and willingness of people to learn and practice CPR and AED by utilizing questionnaires, and then to evaluate the effect of the creative program, which was modified according to the results of the questionnaires, on the motivations and willingness of people to learn and practice CPR and AED.

The investigators expect to design a more efficient resuscitation skill training course by implementing the research project and further to improve the motivations and willingness of people to learn and practice CPR and AED in the future.

ELIGIBILITY:
Inclusion Criteria:

* healthy laypersons without CPR training within two years

Exclusion Criteria:

* non

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
chest compression rate | immediately after the training course
  differences of chest compression rates
chest compression depth | immediately after the training course
  differences of chest compression depth
hands-off time of chest compression | immediately after the training course
  differences of hands-off time of chest compression
score of checklist | immediately after the training course
  differences of scores of checklists

SECONDARY OUTCOMES:
score of satisfaction questionnaire | immediately after the training course
  differences of scores of satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan